CLINICAL TRIAL: NCT04314934
Title: Open Label Extension Study for Patients With Early Alzheimer's Disease (AD) Enrolled in Study ANAVEX2-73-AD-004
Brief Title: OLE of Phase 2b/3 Study ANAVEX2-73-AD-004
Acronym: ATTENTION-AD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Anavex Life Sciences Corp. (Industry)
Collaborators: Anavex Australia Pty Ltd. (Industry); Anavex Germany GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANAVEX2-73-AD-EP-004
Record Dates: First submitted 2019-12-12; First posted 2020-03-19 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — tetrahydro-N, N-dimethyl-2,2-diphenyl-3-furanmethanamine hydrochloride

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active (Experimental): ANAVEX2-73
  Interventions: Drug: ANAVEX2-73

INTERVENTIONS:
Drug: ANAVEX2-73 — Oral capsules
  Other Names: Blarcamesine

SUMMARY:
This is a Phase 2b/3 open-label extension study to evaluate the effects of ANAVEX2-73 on safety and effficacy of daily treatment.

DETAILED DESCRIPTION:
This is a Phase 2b/3 open-label extension study to evaluate the effects of ANAVEX2-73 on safety and effficacy of daily treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previous completion of participation in the ANAVEX2-73-AD-004 double-blind study.
* Participants may be either outpatients, or residents of an assisted-living facility.
* Participants must have a designated study partner, who spends at least 10hrs per week with the participant, in order that assessments e.g. carer burden instruments are completed with true knowledge of the participant.
* No suicidal ideation of type 4 or 5 in the Columbia Suicide Severity Rating Scale (C-SSRS) in the past 3 months (i.e. active suicidal thought(s) with intent but without specific plan, or active suicidal thought(s) with plan and intent) OR suicidal behavior in the past 2 years (i.e. actual attempt, interrupted attempt, aborted attempt, or preparatory acts or behavior).
* Confirmation from the participant that, if of childbearing potential is not pregnant through urine pregnancy testing.

Exclusion Criteria:

* Adverse events (AEs) from the previous study (ANAVEX2-73-AD-004) that have not resolved, are moderate or severe, judged to be possibly related or related to study drug, and considered by the investigator to be a contraindication to extension study participation
* Any condition or laboratory abnormality that would make the subject, in the judgment of the investigator, unsuitable for the study
* Significant history of drug addiction (with the exception of nicotine dependence) or abuse (including alcohol, as defined in DSM-V or in the opinion of the investigator) within the last two years prior to informed consent, or a positive urine drug screen for cocaine, opioid, phencyclidine (PCP), amphetamine or marijuana at screening. Prescription medication yielding a positive drug screen are acceptable except for tricyclic antidepressants (e.g. Amitriptyline, Amoxapine, Desipramine, (Norpramin) Doxepin, Imipramine (Tofranil), Nortriptyline (Pamelor), Protriptyline (Vivactil), Trimipramine (Surmontil)).
* Any known hypersensitivity to any of the excipients contained in the study drug formulation.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 96 weeks
  To continue assessing the safety and tolerability of ANAVEX2-73

SECONDARY OUTCOMES:
ADAS-Cog (Alzheimer Disease Assessment Scale-Cognition) | 96 weeks
  Change from baseline to week 96 in cognition according to the Alzheimer Disease Assessment Scale-Cognition (ADAS-Cog)
ADCS-ADL (Activities of Daily Living) | 96 weeks
  Change from baseline to week 96 in ability to perform daily activities according to the Alzheimer's Disease Cooperative Study-Activities of Daily Living Scale (ADCS-ADL)

CONTACTS AND LOCATIONS:
Locations (51):
- Australia (23):
  - Central Coast Neurosciences Research, Central Coast, New South Wales
  - Hornsby (Northern Sydney Health), Hornsby, New South Wales
  - Sydney, Hornsby, New South Wales
  - KaRa MINDS, Macquarie Park, New South Wales
  - Sydney, Macquarie Park, New South Wales
  - Sydney, Sydney, New South Wales
  - University of Sydney, Sydney, New South Wales
  - Sydney, Sydney, NEW
  - Gold Coast, Gold Coast, Queensland
  - Gold Coast Memory Disorders Clinic, Southport, Quennsland
  - Adelaide, Adelaide, South Australia
  - Melbourne, Belmont, Victoria
  - Geelong Private Medical Centre, Geelong, Victoria
  - Delmont Private Hospital, Glen Iris, Victoria
  - Hammond Care, Malvern, Victoria
  - Melbourne, Malvern, Victoria
  - Austin Health, Melbourne, Victoria
  - Melbourne, Melbourne, Victoria
  - Melbourne, Melbourne N., Victoria
  - McCusker, Nedlands, Western Australia
  - Melbourne, Delmont
  - Hammond Health, Malvern
  - Melbourne, Melbourne E.
- Canada (5):
  - Healthy Brain Aging Labs Uni of Calgary, Calgary, Alberta
  - Bruyere Continuing Care, Ottawa, Ontario
  - Kawartha Centre, Peterborough, Ontario
  - Bay Crest Health Sciences, Toronto, Ontario
  - Toronto Memory Program, Toronto, Ontario
- Germany (8):
  - University of Ulm, Memory Clinic, Ulm, Baden-Wurttemberg
  - Bayreuth Clinic, Hohe Warte Hospital, Bayreuth, Bavaria
  - Technical University of Munich, School of Medicine, München, Bavaria
  - Central Institute of Mental Health, Mannheim, Hesse
  - Goettingen University Medicine, Clinic for Psychiatry and Psychotherapy, Göttingen, Lower Saxony
  - University Hospital, Bonn, Bonn, North Rhine-Westphalia
  - Clinic for Psychiatry and Psychotherapy, Mainz, Rhineland-Palatinate
  - Charite University Medicine, Berlin
- Netherlands (3):
  - Brain Research Center, 's-Hertogenbosch
  - Brain Research Center, Amsterdam
  - Brain Research Center, Zwolle
- United Kingdom (12):
  - MAC Clinical Research, Teesside, County Teesside
  - Glasgow Memory Clinic, Glasgow, Scotland
  - Cognition Health, Guildford, Surrey
  - MAC Clinical Research, Barnsley
  - MAC Clinical Research, Blackpool
  - MAC Clinical Research, Cannock
  - MAC Clinical Research, Leeds
  - MAC Clinical Research, Liverpool
  - Cognition Health, London
  - Imperial College, London
  - MAC Clinical Research, Manchester
  - Cognition Health, Plymouth

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Macfarlane S, Grimmer T, Teo K, O'Brien TJ, Woodward M, Grunfeld J, Mander A, Brodtmann A, Brew BJ, Morris P, Short C, Kurrle S, Lai R, Bharadwaj S, Drysdale P, Sturm J, Lewis SJG, Barton D, Kalafatis C, Sharif S, Perry R, Mannering N, MacSweeney JE, Pearson S, Evans C, Krishna V, Thompson A, Munisamy M, Bhatt N, Asher A, Connell S, Lynch J, Rutgers SM, Dautzenberg PL, Prins N, Oschmann P, Frolich L, Tacik P, Peters O, Wiltfang J, Henri-Bhargava A, Smith E, Pasternak S, Frank A, Chertkow H, Ingram J, Hsiung GR, Brittain R, Tartaglia C, Cohen S, Villa LM, Gordon E, Jubault T, Guizard N, Tucker A, Kaufmann WE, Jin K, Chezem WR, Missling CU, Sabbagh MN. Blarcamesine for the treatment of Early Alzheimer's Disease: Results from the ANAVEX2-73-AD-004 Phase IIB/III trial. J Prev Alzheimers Dis. 2025 Jan;12(1):100016. doi: 10.1016/j.tjpad.2024.100016. Epub 2025 Jan 1. PMID 39800452